CLINICAL TRIAL: NCT05193292
Title: Camrelizumab Combined With Trastuzumab and Chemotherapy in Patients With HER2-positive Advanced Colorectal Cancer: A Prospective, Single-arm, Open-label Study
Brief Title: Camrelizumab Combined With Trastuzumab and Chemotherapy in Patients With HER2-positive Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-CamreTrastumCRC
Record Dates: First submitted 2021-12-12; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Neoplasms; Intestinal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms | interventions — camrelizumab; Trastuzumab; XELOX

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combined with trastuzumab and chemotherapy (Experimental): Camrelizumab: 200mg, iv, 21d for a treatment cycle Trastuzumab: 8 mg/kg loading dose, followed by 6 mg/kg maintenance, iv, 21d for a treatment cycle Chemotherapy will either be XELOX, mFOLFOX6, FOLFIRI, mXELIRI or mIRIS
  Interventions: Drug: Camrelizumab; Drug: Trastuzumab; Drug: XELOX regimen; Drug: mFOLFOX6 regimen; Drug: FOLFIRI regimen; Drug: mXELIRI regimen; Drug: mIRIS regimen

INTERVENTIONS:
Drug: Camrelizumab — 200mg, iv, 21d for a treatment cycle
Drug: Trastuzumab — 8 mg/kg loading dose, followed by 6 mg/kg maintenance, iv, 21d for a treatment cycle
Drug: XELOX regimen — Oxaliplatin, 130 mg/m2, iv, d1; Capecitabine, 1000 mg/m2, po, bid, d1-d14; q3w
Drug: mFOLFOX6 regimen — Oxaliplatin, 85 mg/m2, iv, d1; Leucovorin, 400 mg/m2, iv, d1; 5-FU, 400mg/m2, iv, d1 followed by 1200 mg/(m2·d)*2d, civ, 46h; q2w
Drug: FOLFIRI regimen — Irinotecan, 180 mg/m2, iv, d1; Leucovorin, 400 mg/m2, iv, d1; 5-FU, 400mg/m2, iv, d1 followed by 1200 mg/(m2·d)*2d, civ, 46h; q2w
Drug: mXELIRI regimen — Irinotecan, 200 mg/m2, iv, d1; capecitabine, 800 mg/m2, po, bid, d1-d14; q3w
Drug: mIRIS regimen — Irinotecan, 180 mg/m2, iv, d1; Tiggio Capsules (S-1), 40-60 mg/m2, po, bid, d1-d9; q2w

SUMMARY:
This study aimed to evaluate the efficacy and safety of camrelizumab combined with trastuzumab and chemotherapy in Patients with HER2-positive advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects has voluntarily agreed to sign the informed consent and have good compliance and are willing to cooperate with follow-up.
2. Age 18 years or older, male or female.
3. Have a life expectancy of at least 3 months.
4. Histologically confirmed diagnosis of unresectable recurrent or metastatic HER2 positive colorectal cancer.
5. HER2 positivity defined as the colorectal cancer-specific HERACLES diagnostic criteria or NGS sequencing of tumor tissue/blood samples showed HER2 amplification.
6. Patients have not received systemic anti-cancer treatment in the past or had disease progression more than 6 months after receiving after (neo)adjuvant treatment could be enrolled or failure of first-line therapy or completion of (new) adjuvant therapy to disease recurrence less than 6 months.
7. At least one measurable or evaluable lesion, as defined by RECIST 1.1 criteria.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. The functional level of the major organs must meet the following requirements:(1)Blood routine: neutrophils (ANC) ≥1.5×10^9/L; platelet count (PLT)≥90×10^9/L; hemoglobin (Hb) ≥90 g/L; (2)Blood biochemistry: TBIL≤1.5×ULN; ALT and AST≤2.5×ULN; Cr≤1.5×ULN and creatinine clearance≥50 mL/min (Cockcroft-Gault formula); for subjects with liver metastasis: TBIL≤3×ULN; ALT and AST≤5×ULN; (3)Patients was not receiving anticoagulation therapy (INR ≤ 1.5 or aPTT ≤ 1.5 × ULN). If the patient received prophylactic anticoagulation therapy and the INR ≤ 2 × ULN within 14 days before the start of the study and the aPTT/PPT is within the normal range could be enrolled; (4)Left ventricular ejection fraction (LVEF) ≥55% (within 28 days).
10. Female subjects of childbearing age or male subjects whose sexual partners are females of childbearing age must take effective contraceptive measures throughout the treatment period and 6 months after the treatment period.

Exclusion Criteria:

1. Have previously received any co-stimulatory or co-inhibitory T cell receptor antibody or drug therapy, including PD-1, PD-L1, PD-L2, CD137, CTLA-4, etc.
2. Have previously received anti-HER2 targeted therapy (monoclonal antibody or small molecule TKI).
3. Have any active autoimmune diseases or autoimmune diseases in the past 2 years.
4. Have used immunosuppressive drugs within 4 weeks before the first dose of study drug treatment.
5. Allergic to any monoclonal antibody or chemotherapeutic drug preparation component.
6. Receive a live attenuated vaccine within 4 weeks before the first dose of study drug treatment.
7. Known symptomatic central nervous system metastases and/or cancerous meningitis. If subjects with brain metastases who have been treated in the past are in stable condition, they could be enrolled.
8. Pleural and abdominal effusion requiring clinical treatment, or third interspace effusion.
9. Suffering from congenital or acquired immune deficiency.
10. Known history of human immunodeficiency virus (HIV) infection.
11. Subjects who have received allogeneic tissue/solid organ transplantation.
12. Known to have active tuberculosis.
13. Known to have acute or chronic active hepatitis B or acute or chronic active hepatitis C.
14. Severe infections that are active or poorly clinical controlled.
15. Known history of (non-infectious) pneumonia requiring steroid treatment or currently suffering from pneumonia.
16. Other poorly controlled comorbidities.
17. Pregnancy or breastfeeding or planning to pregnancy or childbirth during the study period.
18. Have uncontrolled cardiac clinical symptoms or diseases.
19. Malignant tumors that are progressing or require active treatment in the past 5 years, except for the following: (1) Malignant tumors that have been completely relieved for at least 2 years before enrollment and no other treatment is required during the study period; (2) Non-melanoma skin cancer or malignant freckle-like nevus that has been adequately treated and has no evidence of disease recurrence; (3) Carcinoma in situ with adequate treatment and no evidence of disease recurrence.
20. According to the judgment of the investigator, the patient has other factors that may affect the results of the study or cause the study to be terminated halfway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | [ Time Frame: Approximately 24 months ]
  The proportion of patients with complete response or partial response according to RECIST v1.1

SECONDARY OUTCOMES:
Progression-Free Survival | [ Time Frame: Approximately 24 months ]
  Time from the initiation of treatment to disease progression or any-cause death
Disease Control Rate | [ Time Frame: Approximately 24 months ]
  The proportion of patients with complete response, partial response or stable disease according to RECIST v1.1
Overall Survival | [ Time Frame: Approximately 24 months ]
  Time from the initiation of treatment to any-cause death
Duration of Response | [ Time Frame: Approximately 24 months ]
  Time from complete response or partial response to disease progression or any-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China